CLINICAL TRIAL: NCT01786239
Title: Detecting Which Patients With Schizophrenia Will Improve With Omega-3 Treatment
Brief Title: Omega-3 Dietary Supplements in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delbert Robinson (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor-Investigator, Delbert Robinson, Psychiatrist, Northwell Health
Organization: Northwell Health (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-308B
Record Dates: First submitted 2013-01-14; First posted 2013-02-07 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Schizophrenia; Schizophreniform Disorder; Schizoaffective Disorder; Bipolar Disorder; Psychosis NOS
Keywords: Adolescence; Adult; Antipsychotic Agents; Female; Human; Male; Risperidone; Omega-3; Schizophrenia; Schizophreniform; Schizoaffective; Schizophrenia -- *drug therapy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Mental Disorders | interventions — Risperidone; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 capsules & Risperidone (Experimental): Subjects will take 1 capsule in the morning and 1 capsule in the evening. Each capsule contains 370 mg EPA and 200 mg DHA as well as 2 mg/g tocopherol. The study dose will start on day 1 and remain the same throughout the study.
  Interventions: Drug: Risperidone; Drug: Omega-3 capsules
- Placebo & Risperidone (Other): Subjects will take 1 capsule in the morning and 1 capsule in the evening.The placebo is a soybean/corn blend (each capsule contains 1000 mg). The study dose will start on day 1 and remain the same throughout the study.
  Interventions: Drug: Risperidone; Drug: Placebo

INTERVENTIONS:
Drug: Risperidone — The dosage for risperidone will be 1 mg to 6 mg per day. The dose of the risperidone will be based on the participant's clinical improvement and side effects.
  Other Names: Risperdal
Drug: Omega-3 capsules — The total daily dose for omega-3 subjects will be 740 mg of eicosapentanoic acid (EPA)and 400 mg of docosahexaenoic acid(DHA). This dose will start on day 1 and stay the same dose until study completion.
  Other Names: Omega-3
  Arms: Omega-3 capsules & Risperidone
Drug: Placebo — The total daily dose for subjects assigned to placebo will be 2000 mg. This dose will start on day 1 and stay the same dose until study completion.
  Other Names: Placebo capsules
  Arms: Placebo & Risperidone

SUMMARY:
This 16-week placebo-control study looks to investigate whether patients with schizophrenia for two years or less may benefit from omega-3 supplements.

DETAILED DESCRIPTION:
This study looks to investigate whether patients with schizophrenia for 2 years or less may benefit from omega-3 supplements. The main hypothesis to be tested in this study is that white matter integrity assessed with diffusion tensor imaging (DTI) and erythrocyte membrane omega-3 concentration may provide the means for identifying patients most likely to derive clinical benefit from omega-3 supplementation.

To test this hypothesis the investigators will enroll 58 patients with recent-onset schizophrenia into a 16-week long randomized double blind placebo-controlled study of risperidone versus risperidone plus omega-3 supplementation. Study assessments after consent will include a baseline MRI and an MRI at the final visit, blood-work, clinical interviews to assess symptoms, and medical assessments for side effects. DTI exams and peripheral omega-3 concentration will be obtained prior to the initiation of treatment and the primary outcome measure will be the total Brief Psychiatric Rating Scale Score.

Specific aims are:

* To examine the efficacy of omega-3 fatty acids as an adjuvant agent in the treatment of patients with recent-onset schizophrenia. The investigators hypothesize that patients treated with omega-3 fatty acids will demonstrate greater Brief Psychiatric Rating Scale (BPRS) reductions compared to the placebo group.
* To identify whether pre-treatment fractional anisotropy (FA) assessed by DTI predicts which patients will derive clinical benefit from omega-3 fatty acids. The investigators hypothesize that patients with lower fractional anisotropy will derive greater clinical benefit from omega-3 fatty acid supplementation.
* To identify whether pre-treatment peripheral omega-3 fatty acid concentrations predict which patients will derive clinical benefit from omega-3 fatty acids. The investigators hypothesize that patients with lower peripheral omega-3 fatty acid concentrations will derive greater clinical benefit from omega-3 fatty acid supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Current DSM-IV-defined diagnosis of schizophrenia, schizophreniform, schizoaffective disorder, psychosis NOS or Bipolar I as assessed using the Structured Clinical Interview for Axis I DSM-IV Disorders;
* Does not DSM-IV criteria for a current substance-induced psychotic disorder, a psychotic disorder due to a general medical condition, delusional disorder, brief psychotic disorder, shared psychotic disorder, or a mood disorder with psychotic features;
* current positive symptoms rated more than 4 (moderate) on one of these BPRS items: conceptual disorganization, grandiosity, hallucinatory behavior, and unusual thought content;
* is in a early phase of illness as defined by having taken antipsychotic medications for a cumulative lifetime period of 2 years or less;
* age 15 to 40;
* competent and willing to sign informed consent; and
* for women, negative pregnancy test and agreement to use a medically accepted birth control method.

Exclusion Criteria:

* serious neurological or endocrine disorder or any medical condition or treatment known to affect the brain;
* any medical condition which requires treatment with a medication with psychotropic effects;
* significant risk of suicidal or homicidal behavior;
* cognitive or language limitations, or any other factor that would preclude subjects providing informed consent;
* medical contraindications to treatment with risperidone (e.g. neuroleptic malignant syndrome with prior risperidone exposure), omega-3 supplements (e.g. bleeding disorder, seafood allergies) or placebo capsules (e.g. allergies to capsule components);
* contraindications to MRI imaging (e.g. presence of a pacemaker);
* lack of response to a prior adequate trial of risperidone;
* taking omega-3 supplements within the past 8 weeks, and
* requires treatment with an antidepressant or mood stabilizing medication.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Delbert G Robinson, MD, Principal Investigator — The Zucker Hillside Hospital
Locations (1):
- The Zucker Hillside Hospital, Glen Oaks, New York, United States

REFERENCES:
- [Derived] Robinson DG, Gallego JA, John M, Hanna LA, Zhang JP, Birnbaum ML, Greenberg J, Naraine M, Peters BD, McNamara RK, Malhotra AK, Szeszko PR. A potential role for adjunctive omega-3 polyunsaturated fatty acids for depression and anxiety symptoms in recent onset psychosis: Results from a 16 week randomized placebo-controlled trial for participants concurrently treated with risperidone. Schizophr Res. 2019 Feb;204:295-303. doi: 10.1016/j.schres.2018.09.006. Epub 2018 Sep 19. PMID 30241990

RESULTS

PARTICIPANT FLOW:
Groups:
- Amber50/50 Soybean Corn Placebo & Risperidone: Subjects will take 1 capsule in the morning and 1 capsule in the evening.The placebo is a soybean/corn blend (each capsule contains 1000 mg). The study dose will start on day 1 and remain the same throughout the study.
  Risperidone: The dosage for risperidone will be 1 mg to 6 mg per day. The dose of the risperidone will be based on the participant's clinical improvement and side effects.
  Amber 50/50 Soybean/Corn Placebo: The total daily dose for subjects assigned to placebo will be 2000 mg. This dose will start on day 1 and stay the same dose until study completion.
Period: Overall Study
Arm/Group | Omega-3 Capsules & Risperidone | Amber50/50 Soybean Corn Placebo & Risperidone
Started | 25 | 25
Completed | 14 | 14
Not Completed | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 Capsules & Risperidone | Placebo & Risperidone | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 25 | 24 | 49
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 18 | 18 | 36
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Structured Clinical interview for DMS-IV (SCID) [Number; unit: participants]
  Schizophreriform | 5 | 5 | 10
  Schizophrenia | 17 | 17 | 34
  Bipolar 1 Disorder | 2 | 2 | 4
  Psychosis NOS | 0 | 1 | 1
  Schizoaffective Disorder | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response
Description: The primary outcome measure will be the total Brief Psychiatric Rating Scale Score. The range of the BPRS is 0 to 126 with higher scores indicated more psychological symptoms.
Time Frame: 16 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Omega-3 Capsules & Risperidone | Placebo & Risperidone
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline BPRS Score | 41.64 (1.44) | 42.38 (1.56)
  Week 16 BPRS Score | 22.5868 (2.1744) | 27.2235 (2.4397)
Statistical Analysis 1: Comparison: Omega-3 Capsules & Risperidone vs Placebo & Risperidone; Test type: Superiority or Other; p = 0.0493, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed throughout the duration of the study. Typically these were assessed at each study visit starting at visit 1-through visits 16.Through study completion up to 16 weeks.
Arm/Group | Omega-3 Capsules & Risperidone | Placebo & Risperidone
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes